CLINICAL TRIAL: NCT00610974
Title: Enhancing Walking in People With Incomplete Spinal Cord Injury by Improving Swing Phase Activity: a Pilot Study
Brief Title: Enhancing Walking in People With Incomplete Spinal Cord Injury: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H07-01394
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Motor-incomplete Spinal Cord Injury
Keywords: Spinal cord injury; walking; gait training; body-weight supported treadmill training; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): One of 2 types of body-weight supported treadmill training (BWSTT) with the Lokomat, which differ only in the level of assistance that the Lokomat provides to leg movements while walking.
  Interventions: Behavioral: Body-weight supported treadmill training
- 2 (Experimental): One of 2 types of body-weight supported treadmill training (BWSTT) with the Lokomat, which differ only in the level of assistance that the Lokomat provides to leg movements while walking.
  Interventions: Behavioral: Body-weight supported treadmill training

INTERVENTIONS:
Behavioral: Body-weight supported treadmill training — BWSTT for 3 times/week for 12 weeks. Each session, subjects will first complete a 10-minute warm-up period followed by 45 minutes of the assigned therapy. Rest breaks will be provided as needed, but subjects must complete 45 minutes of walking per session.
  Arms: 1
Behavioral: Body-weight supported treadmill training — BWSTT for 3 times/week for 12 weeks. Each session, subjects will first complete a 10-minute warm-up period followed by 45 minutes of the assigned therapy. Rest breaks will be provided as needed, but subjects must complete 45 minutes of walking per session.
  Arms: 2

SUMMARY:
The research proposed here will determine the effect of a novel treadmill gait training strategy using a robotic gait trainer (the Lokomat) on functional ambulation in people with SCI. The effect of the new therapy will be evaluated by analyzing changes in functional ambulation and gait patterns during walking.

DETAILED DESCRIPTION:
Community-dwelling individuals with motor-incomplete spinal cord injury will be recruited. In total, 20 participants will be recruited and randomly assigned to one of 2 types of body-weight supported treadmill training (BWSTT) with the Lokomat, which differ only in the level of assistance that the Lokomat provides to the leg movements while walking. Therapy for both groups will take place 3 times/week for 12 weeks. During each session, participants will first complete a 10-minute warm-up period followed by 45 minutes of the assigned therapy. Rest breaks will be provided as needed, but participants should complete 45 minutes of walking per session.

ELIGIBILITY:
Inclusion Criteria:

1. motor-incomplete SCI due to non-progressive lesion (e.g. trauma, ischemia) at least 12 months ago
2. 19 to 65 years of age
3. use of standing or walking as part of typical activities of daily living
4. controlled spasticity (stable administration of anti-spasticity medication) for the duration of the study

Exclusion Criteria:

1. lesion below 11th thoracic level (lower motoneuron injury)
2. weight greater than 300 lbs or height greater than 6'1"
3. femur length <35 cm or >47 cm and body weight >150 kg
4. cardiac, musculoskeletal, or other uncontrolled health condition (e.g. orthostatic hypotension, osteoporosis) for which exercise or treadmill activity is contra-indicated
5. existing skin irritation or open wounds/sores in lower extremity areas in contact with the leg cuffs of the Lokomat or body weight support harness
6. existing cognitive impairment (as indicated by a Cognitive Capacity Screening Examination (CCSE) score of less than 24 out of 30)
7. participation in rehabilitation therapy or other research study with exercise or mobility outcomes

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome is functional ambulation measured before, after, 1-month after, and 6-months after training. | 6 months

SECONDARY OUTCOMES:
Average activity level per day measured before, after, 1-month after, and 6-months after training | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tania Lam, Ph.D, Principal Investigator — University of British Columbia; Janice J. Eng, Ph.D, Study Director — University of British Columbia
Locations (1):
- Human Locomotion Lab, University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Lam T, Pauhl K, Ferguson A, Malik RN; BKin; Krassioukov A, Eng JJ. Training with robot-applied resistance in people with motor-incomplete spinal cord injury: Pilot study. J Rehabil Res Dev. 2015;52(1):113-29. doi: 10.1682/JRRD.2014.03.0090. PMID 26230667